CLINICAL TRIAL: NCT03411070
Title: Using Radar Technology to Tag Abnormal Lymph Nodes for Removal During Surgery Following Neoadjuvant Chemotherapy
Brief Title: SCOUT Reflector for Tagging Lymph Nodes for Targeted Removal in Patients With Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Faxitron bioptics, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-001864; NCI-2017-02394 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-01

CONDITIONS: Positive Axillary Lymph Node; Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (SCOUT reflector surgery) (Experimental): Patients undergo image-guided placement of the SCOUT reflector prior to course 2 of standard of care neoadjuvant chemotherapy. Patients undergo standard of care surgery approximately 4-8 weeks after chemotherapy completion.
  Interventions: Device: Implanted Medical Device; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Device: Implanted Medical Device — Undergo SCOUT reflector placement
  Other Names: IMPLANTED
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This pilot clinical trial will evaluate whether the SCOUT reflector can be used to tag abnormal lymph nodes in patients with breast cancer prior to chemotherapy for targeted removal at the time of surgery. The SCOUT localization system with the SAVI reflector is non-radioactive and completely internal so can be placed into an abnormal lymph node prior to chemotherapy treatment, which theoretically will allow easier identification and therefore more reliable targeting of the abnormal lymph node for surgical removal.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Percentage of patients with successful retrieval of the reflector confirmed by specimen radiography.

II. Percentage of patients with successful retrieval of the biopsied node, confirmed by presence of clip, biopsy changes or treatment-related changes on pathology.

SECONDARY OBJECTIVES:

I. Total number of lymph nodes removed. II. Percentage of patients in which clipped node was a sentinel node. III. Percentage of patients with nodal pathologic complete response (PCR). IV. Residual cancer burden (RCB) score for patients with residual nodal disease.

V. Percentage of patients requiring axillary dissection. VI. Days prior to surgery of reflector insertion.

OUTLINE:

Patients undergo image-guided placement of the SCOUT reflector prior to course 2 of standard of care neoadjuvant chemotherapy. Patients undergo standard of care surgery approximately 4-8 weeks after chemotherapy completion.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent to participate in the study
* Patients with a breast cancer diagnosis of any subtype and a biopsy-proven positive axillary lymph node who will be treated first with chemotherapy
* Enlarged lymph node and/or clip targetable with image guidance
* Patients who are eligible for surgical resection of the primary breast cancer and targeted dissection of the axilla

Exclusion Criteria:

* More than 3 positive axillary nodes on imaging or matted nodes on clinical exam
* Stage IV breast cancer
* Pregnant or lactating females
* Patients with inflammatory breast cancer
* Patients with allergies to isosulfan blue or technetium, which would preclude sentinel node mapping
* Patients who have had previous axillary surgery, including sentinel lymph node biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with successful retrieval of reflector confirmed by specimen radiography | Up to 2 years
Percentage of patients with successful retrieval of the biopsied node, confirmed by presence of clip, biopsy changes or treatment-related changes on pathology | Up to 2 years

SECONDARY OUTCOMES:
Total number of lymph nodes removed | Up to 2 years
Percentage of patients in which clipped node was a sentinel node | Up to 2 years
Percentage of patients with nodal pathologic complete response (PCR) | Up to 2 years
Residual cancer burden (RCB) score for patients with residual nodal disease | Up to 2 years
Percentage of patients requiring axillary dissection | Up to 2 years
Days prior to surgery of tag insertion | Up to 2 years
Incidence of adverse events | Up to 2 years
  All adverse events due to these procedures will be recorded and reported to the institutional review board (IRB).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Baker, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Baker JL, Haji F, Kusske AM, Fischer CP, Hoyt AC, Thompson CK, Lee MK, Attai D, DiNome ML. SAVI SCOUT(R) localization of metastatic axillary lymph node prior to neoadjuvant chemotherapy for targeted axillary dissection: a pilot study. Breast Cancer Res Treat. 2022 Jan;191(1):107-114. doi: 10.1007/s10549-021-06416-z. Epub 2021 Oct 15. PMID 34652548